CLINICAL TRIAL: NCT06411626
Title: Home Reported Outcomes in PNH: A Mobile App-Based, Prospective, Observational Program to Evaluate Disease Burden and Treatment Patterns in Paroxysmal Nocturnal Hemoglobinuria in the US
Brief Title: Home Reported Outcomes in PNH
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLNP023C1US01
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: Paroxysmal nocturnal hemoglobinuria; PNH; home reported outcomes; HRO; patient-reported outcome; PRO; real-world data; iptacopan
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Participants with PNH: Participants with PNH
  Interventions: Other: PNH-relevant therapies

INTERVENTIONS:
Other: PNH-relevant therapies — This is an observational study. There is no treatment allocation. The decision to initiate PNH-relevant therapies (such as eculizumab, ravulizumab, pegcetacoplan, iptacopan, and others) will be based solely on clinical judgement.

SUMMARY:
The study aims to longitudinally capture the full spectrum of symptoms, treatment utilization, and overall Health-Related Quality of Life (HRQoL) experienced by PNH patients. By primarily utilizing home reported outcomes (HRO) data on symptom burden and treatment usage, supplemented with patient-reported outcome (PRO) measures, the study seeks to establish a new real-world data (RWD) source to understand symptom variability and HRQoL among PNH patients, including those receiving orally administered iptacopan.

DETAILED DESCRIPTION:
The study will be prospective and observational, conducted over an initial period of six months per individual from the point of study enrollment. Participants will utilize the Folia mobile app to enroll, consent, and complete all study activities. A hybrid recruitment method of clinic referrals and community referrals will be employed to identify participants, who will be asked to track routine treatment, symptoms, changes in treatment plans, and HRQoL using the Folia Health mobile app. Monthly survey check-ins will be conducted to capture additional data inputs, with the possibility of integrating electronic health record (EHR) and/or claims data.

ELIGIBILITY:
Inclusion Criteria:

Study participants eligible for inclusion in this study must meet all of the following criteria:

* Aged 18 or older
* US-based with a proficient understanding of and ability to read the English language
* Any patient with a diagnosis of PNH, regardless of symptom or treatment history

Exclusion Criteria:

Study participants who do not fit all inclusion criteria listed above are unable to participate in this study. Outside of required inclusion criteria, there are no other exclusion criteria in order to meet the exploratory nature of the primary endpoint.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18+ who have been diagnosed with PNH, regardless of symptom or treatment history, and are US-based with a proficient understanding of and ability to read the English language.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
PNH symptom burden | Baseline, month 6
  Primary endpoint will be measured through longitudinal Home Reported Outcomes (HRO) tracking of self-selected symptoms at enrollment and associated changes in severity against self-reported baselines.

SECONDARY OUTCOMES:
Number of participants by treatment utilization and management of potential flare events | Up to 6 months
  Treatment utilization and management of potential flare events tracked during the study period
Number of participants by reported treatment use and treatment switching | Up to 6 months
  HRO-reported treatment use and treatment switching throughout the study duration, triangulated with symptoms reported throughout the study duration
Health-related quality of life (HRQoL) | up to 6 months
  HRQoL HRO tracking data:
  * Mood & behavioral health
  * Productivity
  * Reasons for discontinuing or changing a treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No